CLINICAL TRIAL: NCT01523314
Title: Topical Dexamethasone - Cyclodextrin Microparticle Eye Drops for Diabetic Macular Edema
Acronym: DECEDE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Ahmed Abu El-Asrar, Professor, Consultant, Vitreoretinal/Uveitis division, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DECEDE
Record Dates: First submitted 2012-01-28; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; intravitreal injection; dexamethasone; Cyclodextrin; eye drops; bevacizumab; macular laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexamethasone - Cyclodextrin (Experimental)
  Interventions: Drug: dexamethasone - Cyclodextrin eye drops
- Avastin/Laser (Active Comparator)
  Interventions: Other: intravitreal Avastin injection +/- macular laser

INTERVENTIONS:
Drug: dexamethasone - Cyclodextrin eye drops — The study eye will receive the dexamethasone NP eye drops 3 times a day for 3 months. The subject will be handed an eye drop bottle at each monthly visit for self administration of the eye drops. Each eye drop container is to be marked with a date when first opened and discarded after 1 week (unless it contains a preservative).
  Arms: dexamethasone - Cyclodextrin
Other: intravitreal Avastin injection +/- macular laser — The study eye will receive standard laser and intravitreal injections of Avastin for 3 months. Complete eye examination will be performed prior to drug administration.
  Arms: Avastin/Laser

SUMMARY:
The research group has developed new ocular drug delivery technology based on cyclodextrin nanoparticles (NP). The investigators plan to develop and test this technology to help treat diabetic macular edema (DME).

An important step in research was the invention of cyclodextrin nanoparticles, which has just received a US patent. The investigators pre-clinical and clinical work has demonstrated the investigators eye drop suspension with cyclodextrin nano-particles to be superior to conventional eye drops. They increase drug absorbance into the eye and decrease systematic distribution of the drug, hence reducing side effects. Cyclodextrin nanoparticle eye drops deliver drugs to the posterior part of the eye, thus solving one of the biggest obstacles in ocular pharmacology.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Pseudophakic in study eye, i.e. with IOL (intra ocular lens) after cataract surgery
* Diabetic macular edema with central macular thickness over 300 µm on OCT in study eye. If both eyes have DME, then the treatment will be applied to the eye with thicker central macula on OCT.
* Age 18 years or older

Exclusion Criteria:

* Glaucoma or use of any glaucoma medication
* Known steroid IOP response
* Any infectious eye disease
* Treatment for DME within 6 months, such as laser treatment, intravitreal or subtenon injections of steroids, intravitreal injections of anti vascular endothelelial growth factor medication.
* Any eye surgery within 3 months or other eye conditions e.g. corneal disorders, ocular hypotony and retinal detachments.
* Crystalline lens present in study eye
* Known allergy to cyclodextrins, dexamethasone, ranibizumab or any of the components of the study medications

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-08 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity on ETDRS chart | 3 months

SECONDARY OUTCOMES:
Intraocular pressure (IOP) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine, King Saud University, Riyadh, Riyadh Region, Saudi Arabia